CLINICAL TRIAL: NCT06966973
Title: Pediatric Polysomnography at Home: Feasibility, Quality, and Satisfaction in Normal Children and Children With Neurodevelopmental Disorders
Brief Title: Ambulatory Polysomnography in Neurodiverse Children: Feasibility, Quality, and Satisfaction
Status: Completed | Type: Observational
Sponsor: UPNOS (Other)
Collaborators: Hôpital Raymond Poincaré (Other); AdSalutem Sleep Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-AMBUPED-001
Record Dates: First submitted 2025-03-13; First posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Neurodevelopmental Disorders; Pediatric Sleep Apnea; Periodic Leg Movements, Excessive, Sleep-Related; Polysomnography
Keywords: Home unattended polysomnography; Attention deficit disorder; Attention deficit hyperactivity disorder; Learning disorders
MeSH Terms: conditions — Neurodevelopmental Disorders; Nocturnal Myoclonus Syndrome; Attention Deficit Disorder with Hyperactivity; Learning Disabilities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- All children aged 2 to 17
  Interventions: Other: Polysomnograpy

INTERVENTIONS:
Other: Polysomnograpy — All successive patients who underwent polysomnography

SUMMARY:
Laboratory polysomnography is the gold standard for objective sleep measurement. With hospital waiting times becoming increasingly long, outpatient polysomnography seems a good solution. Children are at greater risk of developing sleep disorders and polysomnography in the hospital laboratory can be a stressful examination for these children and their parents. This can be even more the case in populations of children with neurodevelopmental disorders, such as Attention Deficit Disorder with or without Hyperactivity (ADHD), or dys- learning disorders. Several studies have already demonstrated the feasibility of ambulatory, in a home setting, polysomnography in children. The objective of this study is to demonstrate the acceptability and satisfaction of performing polysomnography at home on a large cohort of children, including children with neurodevelopmental disorders.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive children who underwent a H-PSH
* Age beetween 2 and 17 years old

Exclusion Criteria:

* No signed informed consent form for study participation

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study population consisted of any children coming to the doctor's office for a home unattended polysomnography, aged between 2 and 17 years at the time of polysomnography, and whose parents had signed a consent form for polysomnography and data collection.
Sampling Method: Non-Probability Sample
Enrollment: 563 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Acceptability of Home Unattended Polysomnography | One day after the polysomnography
  Parents and children completed 10 cm visual analog scales (VAS) to assess their satisfaction with the home recording (scored from 0 (not enjoyed) to 10 (very satisfied) and preference for home versus laboratory PSG (scored from 0 preference for H-PSG to 10 preference for L-PSG).

SECONDARY OUTCOMES:
List of symptoms prompting polysomnographic examination | During the polysomnography analysis
  The following symptoms are collected through a standardized questionnaires completed by participants. Only the presence or absence of each symptom is recorded: Disturbed attention; Fatigue;Snoring; Nocturnal sweating; Kick; Enuresis; Nocturnal awakening; Sleepiness PPDS > 16; Morning headache; Difficulty staying asleep.
Global signal quality across all channels of the polysomnographic recording. | One night of polysomnography.
  Global assessment of signal integrity across all polysomnography channels, expressed as a percentage over the course of a full-night recording.
SpO₂ signal quality of the polysomnographic recording. | One night of polysomnography.
  SpO₂ signal quality expressed as a percentage over the course of a full-night recording.
Nasal cannula signal quality of the polysomnography recording. | One night of polysomnography.
  Nasal cannula signal quality expressed as a percentage over the course of a full-night recording.
RIP (Respiratory Inductance Plethysmography) quality of the polysomnography recording. | One night of polysomnography.
  RIP (Respiratory Inductance Plethysmography) quality expressed as a percentage over the course of a full-night recording.
Sleep latency assessed by Polysomnography. | One night of polysomnography.
  Time from lights-off to the onset of sleep in minutes
Sleep Efficiency assessed by Polysomnography. | One night of polysomnography.
  Sleep efficiency=total sleep time/total bed rest time x 100% according to the Polysomnography, expressed as a percentage.
REM latency assessed by Polysomnography. | One night of polysomnography.
  Time from sleep onset to the first epoch of Rapid Eyes Movement (REM) sleep in minutes.
Arousal Index assessed by Polysomnography. | One night of polysomnography.
  Number of electroencephalography arousals per hour of sleep assessed by Polysomnography.
Sleep Stage Distribution assessed by Polysomnography | One night of polysomnography.
  Sleep stage distribution during nocturnal sleep, defined as the percentage of total sleep time spent in N1, N2, N3, and REM stages, assessed by polysomnography
Number of Periodic Limb Movements per Hour of Sleep (PLMS Index), measured by Polysomnography. | One night of polysomnography.
  Number of periodic limb movements per hour of sleep (PLMS Index), assessed by Polysomnographic recording of bilateral anterior tibialis electromyography.
Respiratory events during sleep assessed by Polysomnography | One night of polysomnography.
  Respiratory events during nocturnal sleep. This includes saturation, nasal air flow and movement of the stomach and chest, together showing the number of apneas and hypopneas per hour of sleep assessed by full-night polysomnographic recording.

CONTACTS AND LOCATIONS:
Locations (1):
- UPNOS, Garches, France

IPD SHARING:
Plan to Share IPD: Undecided
Observational study on routine practice. The individual data collected are specific to the protocol and cannot be directly reused without the full set of tools and methodologies developed for this study. Their dissemination could be misinterpreted or non-reproducible outside this context.

REFERENCES:
- See also: Related Info — https://www.health-data-hub.fr/projets/polysomnographie-pediatrique-domicile-acceptabilite-et-satisfaction-chez-des-enfants